CLINICAL TRIAL: NCT04823598
Title: Comparing Spontaneous Versus Interventionist Approaches: A Randomized Controlled Study on the Impact of Manual Perineal Protection and Pushing Techniques on Perineal Outcomes in Nulliparous Women
Brief Title: Pushing and Manual Perineal Protection Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Refika Genc Koyuncu, assistant professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HonHoP
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Perineal Tear; Episiotomy Extended by Laceration; Labor Complication
Keywords: Episiotomy; Obstetric Labor Complications; Perineum
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Active Comparator): Coached pushing and Finnish manual perineal protection
  Interventions: Procedure: Coached pushing and Finnish manual perineal protection
- Study group (Experimental): Uncoached pushing and Hands-poised perineal protection
  Interventions: Procedure: Uncoached pushing and Hands-poised perineal protection

INTERVENTIONS:
Procedure: Coached pushing and Finnish manual perineal protection — Pushing technique: Rest will be encouraged between uterine contractions. With the onset of uterine contraction, women will be instructed to breathe normally. They will then be instructed to take a deep breath and hold (closed-glottis), and push down strongly for as long as possible (up to 10 seconds). After pushing effort, normal breathing will be encouraged, then the same pushing instruction will be repeated again.
  Fetal expulsion: The expulsion rate of the fetal head will be controlled by light pressure applied on the fetal occiput. Simultaneously, the thumb and index finger of the dominant hand will be used to support the perineum, while the bent middle finger will grasp the baby's chin. Once a good grip is achieved, the investigator slowly assists in the expulsion of the fetal head from the vaginal introitus. When most of the fetal head is out, the perineal ring will be pushed under the baby's chin.
  Arms: Reference group
Procedure: Uncoached pushing and Hands-poised perineal protection — Women will not be given any instructions regarding straining and breathing, and will be allowed to follow their own pushing impulses. During the expulsion of the fetal head, the hands of the researcher will be kept in the air and ready for the intervention, but pressure will not be applied to the fetal head or perineum unless necessary (fetal hypoxic appearance, strain detection with a risk of spontaneous laceration towards the anus in the midline).
  Arms: Study group

SUMMARY:
Perineal trauma during vaginal delivery is very common, especially in countries with a high prevalence of episiotomy. Perineal traumas can range from tears limited to the skin, subcutaneous and vaginal mucosa to severe tears involving the anal sphincter and rectal mucosa. Perineal trauma is associated with short-term morbidities such as bleeding, infection, pain, edema. Besides, it may cause long-term morbidities such as urinary incontinence, fecal incontinence, dyspareunia, a decrease in quality of life, a need for surgery, and psychosocial problems. Moreover, it is associated with an increase in national healthcare costs and malpractice cases. For these reasons, some measures to reduce the frequency of perineal trauma have been discussed for many years. Pushing techniques applied in the second stage of labor and manual perineum protection techniques applied during fetal expulsion are among these. Current data are insufficient to make definitive recommendations. In this study, it was aimed to compare different pushing and perineal protection techniques in the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* 37-40 weeks of gestation
* Singleton pregnancy
* Vertex presentation
* Risk-free pregnancy
* Estimated fetal weight 2500-4000 g
* In the first stage of birth
* Amniotic membranes are intact
* Adequate knowledge of written and spoken Turkish

Exclusion Criteria:

* Cesarean delivery need
* Need for labor induction
* Need for operative delivery (vacuum, forceps)
* Need for obstetric analgesia
* Kristaller maneuver
* Perineal preparation during pregnancy (perineal massage in the last month of pregnancy, etc.)
* Vulvo-vaginal infection
* Vulvar severe varicose veins
* Postpartum atony
* Non-compliance with research follow-up criteria
* Covid-19 positivity
* Non-compliance with the procedure of the group involved
* Neuropsychiatric and other diseases that cause understanding, speech, and expression disorders

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nulliparous pregnant women in the first stage of labor will be included in the study.
Enrollment: 164 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Episiotomy | between the end of the second stage of labor and fetal expulsion
  Episiotomy rates
Perineal lacerations | between the end of the second stage of labor and fetal expulsion
  Frequency of perineal lacerations according to their severity

SECONDARY OUTCOMES:
Perineal pain | 24th hour after birth
  Average pain score obtained by the Visual Analog Scale
Maternal birth satisfaction | 24th hour after birth
  Average score obtained by the Birth Satisfaction Scale
Breastfeeding | 24th hour after birth
  Average score obtained by the Bristol Breastfeeding Assessment Tool
Anal incontinence | 1th month after birth
  Mean anal incontinence score obtained by Wexner scale
Pelvic muscle function | 1th month after birth
  Mean scores obtained by the "PERFECT scheme" regarding pelvic floor muscle function (total and subscale scores)

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Genc Koyucu R, Ketenci Gencer F, Bilici SR. Effects of manual perineal protection and pushing techniques used in the second stage of labor on perineal outcomes: a randomized controlled trial of combinations of strategies. BMC Pregnancy Childbirth. 2025 Jun 19;25(1):671. doi: 10.1186/s12884-025-07564-6. PMID 40537769